CLINICAL TRIAL: NCT01168414
Title: A Randomized, Comparison of the Effects of Ganfort and Duotrav on Intraocular Pressure in Patients With Primary Open Angle Glaucoma or Ocular Hypertension Open Label/Evaluator-blind/Cross-over Study
Brief Title: A Study of Ganfort Versus Duotrav in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Dr. Lee Ming Yueh, Ophthalmology Department, Hospital Kuala Lumpur
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-10-466-5929
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Ocular Hypertension; Primary Open Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Ganfort; Duotrav

ARMS (2):
- Ganfort (Active Comparator): Fixed combination of Bimatoprost and Timolol
  Interventions: Drug: Ganfort
- Duotrav (Active Comparator): Fixed combination of Travoprost and Timolol
  Interventions: Drug: Duotrav

INTERVENTIONS:
Drug: Ganfort — Fixed combination of Bimatoprost and Timolol (BTFC; Ganfort (300 microgram + 5 mg/ml eyedrops solution)
  Arms: Ganfort
Drug: Duotrav — Fixed combination of Travoprost and Timolol (TTFC; Duotrav (40 micrograms + 5 mg/ml eyedrops solution)
  Arms: Duotrav

SUMMARY:
This is a single-center, cross-over comparison parallel group randomized trial designed to evaluate the efficacy and safety of Ganfort compared to Duotrav for a treatment period of 8 weeks each.

ELIGIBILITY:
Inclusion Criteria:

1. Visual acuity 6/60 or better
2. Patients who are controlled (IOP < 21 mmHg) on non-fixed combination of Latanoprost & Timolol for at least 3 months before the baseline visit and
3. Patients on mono-therapy either Latanoprost or Timolol who are eligible for dual therapy being not satisfactorily controlled (IOP>21mmHG)

Exclusion Criteria:

1. Angle closure glaucoma
2. Neovascular Galucoma
3. Secondary open angle glaucoma
4. Ocular infection/inflammation within 3 months
5. Ocular surgery within 3 months
6. History of Refractive surgery
7. Argon laser trabeculoplasty/Selective laser trabeculoplasty
8. Pregnancy/nursing
9. Hypersensitivity to benzalkonium chloride or to any other components of the trial drugs solution.
10. Patients in whom beta-blockers are contraindicated
11. Patients on any drugs known to affect IOP.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Mean intraocular pressure of the 12-hour IOP curve | 8 weeks
  To compare the mean intraocular pressure of the 12-hour IOP curve for Ganfort and Duotrav

SECONDARY OUTCOMES:
Mean intraocular pressure | 12 hours
  Difference in mean IOP for Ganfort and Duotrav

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology Department, Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur, Malaysia